CLINICAL TRIAL: NCT06856252
Title: Human Liver ORganoids as a Model to Study the Role of the I148M Variant of the PNPLA3 Gene in the Development of Non-Alcoholic SteatOhepatitis (NASH)
Brief Title: Human Liver ORganoids as a Model to Study the Development of Non-Alcoholic SteatOhepatitis (NASH)
Acronym: REASON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Valenti:, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REASON
Record Dates: First submitted 2024-03-08; First posted 2025-03-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Biospecimen collection of tissue samples from patients undergoing liver resection (both intratumoral and extratumoral tissues in case of hepatocellular carcinoma) or collected from post-transplant whole livers. These samples will allow us to isolate cells (ovalocytes - hepatic progenitor cells) to generate organoids from normal liver tissues (cholecystectomy) and suspected NASH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver resection to isolate cells (Experimental): Isolation and culture of organoids Isolation of hepatic stellate cells Isolation and culture of sinusoidal stellate cells Generation of assembloids
  Interventions: Genetic: Liver resection to isolate cells

INTERVENTIONS:
Genetic: Liver resection to isolate cells — Isolation and culture of organoids Isolation of hepatic stellate cells Isolation and culture of sinusoidal stellate cells Generation of assembloids

SUMMARY:
The primary objective of the study is to generate and characterize three-dimensional models, called "assembloids", composed of the main liver cell populations (in particular from the co-culture of organoids with stellate cells, responsible for fibrogenesis, deriving from clinical samples). These models will be used in order to imitate the first phases of the onset of steatohepatitis, in conditions of altered lipid metabolism (induced through exposure to the main environmental determinants of this condition: excess fatty acids, fructose, cholesterol) in the presence or absence of the mutation I148M of PNPLA3. Other genetic variants will also be analyzed, such as TM6SF2, MBOAT7 and GCKR, which have previously been correlated with the development of non-alcoholic steatohepatitis.

Further objectives will be: 1) identify new biomarkers of pathological activation of human stellate cells and progression of liver damage, to be subsequently validated in clinical case series for future use in clinical management for individual risk stratification; 2) study the epigenetic factors that underlie the onset of non-alcoholic steatohepatitis and its progression to fibrosis, cirrhosis and HCC; 3) evaluate the impact of antisense oligonucleotides directed against PNPLA3 on the severity of the "steatohepatitic" phenotype (lipid accumulation, lipotoxicity and inflammation and fibrogenesis) in assembloids

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) represents the main cause of liver damage and is found in approximately one third of the population (25-30%). NAFLD encompasses a broad spectrum of conditions ranging from simple steatosis to nonalcoholic steatohepatitis (NASH). NASH is found in 20-30% of patients with NAFLD and can progress to cirrhosis and hepatocellular carcinoma.

Progress recorded in recent years in the field of genetics has highlighted how genetic factors play a key role in the susceptibility, severity and long-term prognosis of the disease. In particular, in a genome-wide association study conducted on a multi-ethnic population, the PNPLA3 gene was identified as the main genetic factor that is strongly associated with intra-hepatic fat content, independently of body mass and insulin resistance.

The primary objective of the study is to generate and characterize three-dimensional models, called "assembloids", composed of the main liver cell populations (in particular from the co-culture of organoids with stellate cells, responsible for fibrogenesis, deriving from clinical samples). These models will be used in order to imitate the first phases of the onset of steatohepatitis, in conditions of altered lipid metabolism (induced through exposure to the main environmental determinants of this condition: excess fatty acids, fructose, cholesterol) in the presence or absence of the mutation I148M of PNPLA3. Other genetic variants will also be analyzed, such as TM6SF2, MBOAT7 and GCKR, which have previously been correlated with the development of non-alcoholic steatohepatitis.

Further objectives will be: 1) identify new biomarkers of pathological activation of human stellate cells and progression of liver damage, to be subsequently validated in clinical case series for future use in clinical management for individual risk stratification; 2) study the epigenetic factors that underlie the onset of non-alcoholic steatohepatitis and its progression to fibrosis, cirrhosis and HCC; 3) evaluate the impact of antisense oligonucleotides directed against PNPLA3 on the severity of the "steatohepatitic" phenotype (lipid accumulation, lipotoxicity and inflammation and fibrogenesis) in assembloids

ELIGIBILITY:
Adult patients who have given consent to participate in the study and listed for the following procedures will be included:

* liver biopsy for suspected non-alcoholic steatohepatitis (NASH) at the time of diagnosis;
* liver resection for hepatocarcinoma or other liver lesions (including secondaries from other neoplasms and benign focal lesions, which will allow obtaining healthy starting liver tissue);
* post-transplant healthy liver biopsies;
* cholecystectomies.

It will also be required:

* availability to sign informed consent for the study
* availability of DNA sample for genetic analysis and clinical data,
* blood sampling for genetic and epigenetic analyzes and analysis of non-coding RNAs (lncRNAs, miRNAs and circRNAs).

Patients will be excluded who present:

* positivity for chronic viral hepatitis (HCV-RNA and/or HBsAg);
* positivity to other liver diseases such as autoimmune and viral hepatitis (hepatitis B and C), hereditary hemochromatosis, alpha-1-antitrypsin deficiency, Wilson's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Generation of treatment-related assembloids | up to 35 months
  Isolation of epithelial cells to impact assessment of the I148M variant on the steatohepatic phenotype in human liver assembloids and analysis of the variants of the TM6SF2, MBOAT7 and GCKR genes previously related to the development of non-alcoholic steatohepatitis
Rate of PNPLA3 p.I148M variant in steatohepatitis development through human liver organoids | up to 35 months
  * Knowledge of the gene expression of lipotoxicity and expression of inflammatory markers;
  * Knowledge of the molecular mechanisms to evaluate the state of activation of star cells, the metabolism of retinol and the deposition of extracellular matrix and estimate

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT06856252/Prot_000.pdf